CLINICAL TRIAL: NCT07281859
Title: heaRtInsiGHT Alert guIDE: RightAIDE Application of the HeartInsight Acute Heart Failure Predictor in Routine Clinical Practice: Organizational Models and Workflow.
Acronym: RightAIDE
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: RightAIDE
Record Dates: First submitted 2025-11-26; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Remote Cardiac Monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RightAIDE study is a prospective, multicenter, observational registry designed to evaluate the real-world application of the HeartInsight™ algorithm for predicting acute heart failure (HF) events in patients implanted with a Biotronik ICD or CRT-D device with atrial sensing and Home Monitoring capability. Heart failure is a growing public health issue with high morbidity, mortality, and healthcare costs. HeartInsight, derived and validated in the SELENE HF study, integrates temporal trends of seven physiological variables monitored by the implanted device to provide early warnings of impending acute decompensation, with a median lead time of 42 days. This study aims to collect data on the implementation of a standardized workflow for interpreting and responding to HeartInsight alerts in routine clinical practice. Approximately 100 patients across 14 centers in Italy will be enrolled and followed for 12 months. The primary endpoint is the proportion of HeartInsight alerts considered "actionable," meaning they trigger at least one predefined clinical action (e.g., device reprogramming, therapy optimization, unscheduled visits, or hospital admission). Secondary endpoints include alert frequency, cumulative alert duration, number of patient interviews performed, hospitalizations during and outside alert periods, and the proportion of patients successfully using the HeartInsight Patient App. Data will be collected via electronic case report forms (eCRFs), analyzed descriptively, and monitored for quality. The study will generate insights into integrating HeartInsight-based predictive monitoring into clinical workflows to potentially improve patient management and outcomes.

DETAILED DESCRIPTION:
Study Title:

heaRtInsiGHT Alert guIDE: RightAIDE - Application of the HeartInsight acute heart failure predictor in routine clinical practice, organizational models and workflow

Background and Rationale:

Heart failure is a chronic and progressive condition characterized by the inability of the heart to adequately pump blood to meet the body's needs. It is associated with frequent hospitalizations due to episodes of acute decompensation, which substantially contribute to the burden on healthcare systems.

Recent technological advances have enabled the development of predictive algorithms that analyze remotely transmitted data from implanted cardiac devices to forecast clinical events. HeartInsight™ is an integrated algorithm within Biotronik ICDs and CRT-Ds that evaluates trends in seven key physiological parameters: mean and nocturnal heart rate, atrial high-rate episodes, daily physical activity, heart rate variability, ventricular extrasystoles, and thoracic impedance.

HeartInsight, validated in the SELENE HF study, demonstrated the ability to predict 66 percent of heart failure hospitalizations, providing a median lead time of 42 days. Despite this evidence, prospective real-world data on the integration of HeartInsight within routine clinical practice, supported by a structured clinical workflow, are currently lacking.

Study Design:

RightAIDE is a prospective, multicenter, observational registry designed to evaluate the clinical application of HeartInsight in standard practice. Fourteen Italian centers with expertise in remote monitoring of cardiac implantable devices will participate. Additional centers may be added if needed without constituting a protocol amendment.

Approximately 100 patients will be enrolled and followed for 12 months. Enrollment will be non-consecutive to reflect clinical practice. No investigational procedures or additional diagnostic tests will be required. All devices and software used in this study are CE marked and will be used within their approved indications.

Study Objectives:

The primary objective is to quantify the proportion of HeartInsight alerts that lead to a clinical action. Clinical actions include device reprogramming, reinforcement or optimization of prescribed therapy, unscheduled outpatient visits, additional diagnostic testing, or hospitalization linked to the alert period.

Secondary objectives include evaluating the frequency of alerts, the cumulative duration of alert periods per patient, the number of patient interviews during alert periods, hospitalization rates during and outside alert periods, and the proportion of patients able to install and effectively use the HeartInsight Patient App.

Endpoints:

Primary Endpoint: Percentage of actionable alerts, defined as alerts that result in one or more predefined clinical actions.

Secondary Endpoints: Frequency of alerts per patient, cumulative duration of alert periods, number of telephone interviews conducted in response to alerts, frequency of cardiovascular hospitalizations during and outside alert periods, and rate of Patient App utilization.

Study Procedures:

After verification of eligibility and signing of informed consent, patients will be instructed on the use of the Home Monitoring system, the HeartInsight algorithm, and the optional installation of the Patient App. Patients will be followed for 12 months with remote monitoring and regular clinical visits according to standard care.

When an alert is triggered, the predefined workflow will guide clinical response, including verification of device data, assessment of patient compliance and symptoms, and appropriate interventions as deemed necessary by the treating physician.

Reasons for early withdrawal include interruption of Home Monitoring transmissions for more than 90 days, device removal or replacement, withdrawal of consent, or death.

Sample Size and Statistical Analysis:

Based on prior data from the SELENE HF study indicating an alert rate of approximately 1.1 per patient-year, 91 patients are expected to generate around 100 alerts during the 12-month follow-up. To account for an estimated 10 percent dropout rate, the planned enrollment is 100 patients.

Descriptive statistics will summarize baseline and outcome data. Continuous variables will be reported as quartiles and medians, while categorical variables will be reported as frequencies and percentages. Point estimates and 95 percent confidence intervals will be provided for actionable alert rates and for the incidence of clinical interventions. Statistical analyses will be performed using R software.

Data Management and Confidentiality:

Study data will be collected through electronic case report forms. Personal identifiers will be stored separately from coded study data. Data will be securely stored and retained for up to 15 years in accordance with regulatory requirements.

Ethical Considerations:

The study will be conducted in accordance with the Declaration of Helsinki, Good Clinical Practice (ICH E6 R2), and applicable national regulations. Written informed consent is required prior to participation. Any protocol amendments that could impact patient safety, study endpoints, or key procedures will require ethics committee approval.

Monitoring and Dissemination:

Monitoring will be performed according to a predefined plan to ensure data integrity and protocol compliance. Study results will be disseminated through scientific conferences and peer-reviewed journals. Authorship of publications will be assigned according to predefined performance criteria among participating centers.

Duration:

The enrollment period is planned for approximately 12 months. Each patient will be followed for 12 months, resulting in an overall study duration of approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* The patient has already received a de novo ICD (DR or DX) or CRT-D within no more than one year, according to guidelines, equipped with atrial sensing and a Home Monitoring system.
* Documentation of heart failure of ischemic or non-ischemic origin.
* At the time of device implantation: ejection fraction ≤35% and NYHA Class II or III.
* Sinus rhythm.
* Age ≥18 years.
* The patient has signed the informed consent for participation.

Exclusion Criteria:

* Patients who have received the implantable device as a replacement or upgrade of a previous one.
* Patients who have received the device more than one year ago.
* At the time of enrollment: patient with HeartInsight previously activated.
* Permanent or long-standing atrial fibrillation.
* Sinus node disease with indication for atrial pacing.
* At the time of enrollment: NYHA Class IV.
* Planned cardiac surgery within three months following enrollment.
* Life expectancy of less than one year.
* Unstable residence or insufficient GSM coverage at the patient's home.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with heart failure of ischemic or non-ischemic origin who have been recently implanted with a Biotronik implantable cardioverter defibrillator (ICD) or a cardiac resynchronization therapy defibrillator (CRT-D) with atrial sensing capability and Home Monitoring functionality.
  Eligible patients must have a left ventricular ejection fraction (LVEF) ≤35% and NYHA functional class II or III at the time of device implantation, be in sinus rhythm, and have provided written informed consent.
  Patients are excluded if they have received the device as a replacement or upgrade, have had the device implanted for more than one year, have permanent or long-standing atrial fibrillation, require atrial pacing due to sinus node disease, are in NYHA Class IV, are scheduled for cardiac surgery within three months, have a life expectancy of less than one year, have unstable residence or insufficient GSM coverage for Home Monitoring, or are pregnant or breas
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Actionable alerts | 1 year
  Percentage of actionable alerts, defined as alerts that result in one or more predefined clinical actions.

SECONDARY OUTCOMES:
Frequency of HeartInsight Alerts | 1 year
  Number of HeartInsight alerts generated for each patient during the 12-month follow-up period.
Cumulative Duration of Alert Periods per Patient | 1 year
  Total cumulative duration, in days, of alert periods per patient during the follow-up, considering periods with the recovery threshold active.
Frequency of Telephone Contacts for Patient Interviews | 1 year
  Number of telephone contacts performed with patients during alert periods, as specified in the predefined workflow.
Frequency of Cardiovascular Hospitalizations | 1 year
  Number of hospitalizations for cardiovascular causes during periods of HeartInsight alert and outside alert periods.
Proportion of Patients Using the HeartInsight Patient App | 1 year
  Percentage of patients able to install and effectively use the HeartInsight Patient App during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Dario Gregori, Full Professor, Study Chair — Unit of Biostatistics, Epidemiology and Public Health - UBEP, University of Padova; Gabriele Zanotto, MD, Principal Investigator — Dipartimento di Cardiologia, Ospedale Magalini di Villafranca
Locations (12):
- Italy (12):
  - Clinica Montevergine, Mercogliano, Avellino
  - Spedali Civili di Brescia, Brescia, Brescia
  - Presidio Ospedaliero di Rho - ASST Rhodense, Rho, Milano
  - Ospedale San Gerardo, Monza, Monza
  - Ospedale Monaldi, Napoli, Napoli
  - Ospedale Giovanni Paolo II, Ragusa, Ragusa
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Ospedale Civile SS. Annunziata, Sassari, Sassari
  - Ospedale di Cattinara, Trieste, Trieste
  - Ospedale Mater Salutis di Legnagno, Legnago, Verona
  - Ospedale Fracastoro, San Bonifacio, Verona
  - Ospedale Magalini di Villafranca, Villafranca di Verona, Verona